CLINICAL TRIAL: NCT06651788
Title: Does "Freeze Spray" Work? Evaluating the Efficacy of Ethyl Chloride Usage Prior to Orthopaedic Injections
Brief Title: Does Ethyl Chloride Spray Work?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB23-2039
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-04

CONDITIONS: Injection Fear; Injection Pain Prevention; Injection Complication
Keywords: Injection; Freeze spray; corticosteroid injections; Ethyl chloride; Orthopeadics
MeSH Terms: conditions — Iatrophobia | interventions — Ethyl Chloride

STUDY DESIGN:
Intervention Model Description: the freeze spray group (receiving freeze spray before the injection)
Who Masked: Participant, Care Provider
Masking Description: The study will be double-blinded to minimize bias. After selection into either spray group the cans will be disguised only showing a number 1 or number 2.
  Given that the freeze spray is a skin refrigerant, the saline placebo will be refrigerated to mimic the temperature on the skin. The freeze spray is odorless, as is saline, so should not pose a different in smell experience. Neither the participants or physicians will be unblinded at any point; the unblinded investigator will be the only person with access to unblinded data..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Freeze spray group (Experimental): Ethyl Chloride Usage Prior to Orthopaedic Injections
  Interventions: Other: Ethyl Chloride
- Placebo application of cold saline spray (Placebo Comparator): Saline spray before injection
  Interventions: Other: Cold Saline Spray
- No spray prior to injection (No Intervention): No intervention before injection

INTERVENTIONS:
Other: Ethyl Chloride — Topical anesthetic that rapidly cools the skin and underlying tissues
  Arms: Freeze spray group
Other: Cold Saline Spray — placebo application of cold saline spray
  Arms: Placebo application of cold saline spray

SUMMARY:
A procedure frequently performed by orthopaedic providers is the administration of corticosteroid injections for the management of various soft tissues and joint-related conditions, such as osteoarthritis, tendinitis, carpal tunnel syndrome, trigger finger, and de Quervain's tenosynovitis. While these injections have demonstrated effectiveness in alleviating symptoms, the discomfort associated with the procedure can be a source of anxiety and apprehension for patients. This discomfort arises from the sensation of the needle entering the affected area and the burning sensation induced by the corticosteroid solution.

DETAILED DESCRIPTION:
A procedure frequently performed by orthopaedic providers is the administration of corticosteroid injections for the management of various soft tissues and joint-related conditions, such as osteoarthritis, tendinitis, carpal tunnel syndrome, trigger finger, and de Quervain's tenosynovitis. While these injections have demonstrated effectiveness in alleviating symptoms, the discomfort associated with the procedure can be a source of anxiety and apprehension for patients. This discomfort arises from the sensation of the needle entering the affected area and the burning sensation induced by the corticosteroid solution.

In response to this concern, orthopaedic providers have turned to freeze sprays (Ethyl chloride), which are topical anesthetics that rapidly cool the skin and underlying tissues. By numbing the injection site superficially, freeze sprays offer the potential to mitigate patient discomfort during corticosteroid injections, thus improving the overall patient experience and potentially enhancing treatment compliance.

However, despite the popularity of freeze spray usage in orthopaedics, many orthopaedic providers have concerns about its efficacy when it comes to providing pain relief. There still needs to be comprehensive scientific evidence evaluating its efficacy and safety. A previous study evaluated the efficacy of freeze spray in hand surgery in a randomized study of 150 subjects without standardized outcomes measures. These investigators showed no difference between those receiving freeze spray vs no spray in pain or anxiety; another study of vapocoolant spray in IV start sites in the emergency department similarly showed no difference in pain or anxiety. Based on the literature, there is no definitive standard of care to use freeze spray with injections and this is the gap in knowledge we wish to answer with a rigorous, placebo-controlled study. This study will differ from the previous similar study in that the investigators will recruit double the number of patients and use standardized commonly accepted questionnaires. The use of a questionnaire based on standardized metrics will provide a more comprehensive assessment of patient perceptions and satisfaction with the use of freeze spray. Through a rigorous research approach, the investigators aim to provide valuable insights into the impact of freeze spray on patient comfort, injection success rates, and any potential complications associated with its use.

This study will contribute to the ongoing efforts of hand surgeons to refine their techniques, minimize patient discomfort, and optimize the delivery of corticosteroid injections. Ultimately, the investigators' findings may have significant implications for the broader field of musculoskeletal medicine, offering evidence-based guidance to improve the patient experience and outcomes in orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Receiving a corticosteroid injection in an upper or lower extremity (to include soft tissue and joint injections) for the first time

Exclusion Criteria:

* Patients with previous injection experiences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine if freeze spray usage before corticosteroid injections significantly reduces patient discomfort during the procedure as measured by pain scores before injection | 10 minutes before subject receives injection
  Using the visual analog pain scale (0 no pain - 10 worst possible pain) to ask patients their pain rating and if freeze spray usage before corticosteroid injections significantly reduces patient discomfort during the procedure.
To determine if freeze spray usage before corticosteroid injections significantly reduces patient discomfort during the procedure as measured by pain scores after injeciton | 10 minutes after subject receives injection
  Using the visual analog pain scale (0 no pain - 10 worst possible pain) to ask patients their pain rating and if freeze spray usage before corticosteroid injections significantly reduces patient discomfort during the procedure.
To assess patient perception of freeze spray efficacy in decreasing anxiety regarding injections. | 10 minutes after subject receives injection
  Using the treatment satisfaction questionnaire for medication-II to ask patients their anxiety and if freeze spray usage before corticosteroid injections significantly reduces patient anxiety during the procedure.
To assess their current overall status compared to their pre-injection baseline | 10 minutes after subject receives injection
  Using the single assessment numeric evaluation (0% furthest from normal and 100% normal) to ask patients their current status

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randall DJ, Zhang Y, Li H, Hubbard JC, Kazmers NH. Establishing the Minimal Clinically Important Difference and Substantial Clinical Benefit for the Pain Visual Analog Scale in a Postoperative Hand Surgery Population. J Hand Surg Am. 2022 Jul;47(7):645-653. doi: 10.1016/j.jhsa.2022.03.009. Epub 2022 May 27. PMID 35644742
- [Background] Edwards C, Noah C. A Randomized, Double-Blind Trial to Determine if Vapocoolant in the Adult Population Improves Patient Perception of Pain With Peripheral Intravascular Access. Adv Emerg Nurs J. 2017 Oct/Dec;39(4):288-294. doi: 10.1097/TME.0000000000000165. PMID 29095180
- [Background] Franko OI, Stern PJ. Use and Effectiveness of Ethyl Chloride for Hand Injections. J Hand Surg Am. 2017 Mar;42(3):175-181.e1. doi: 10.1016/j.jhsa.2016.12.013. PMID 28259274
- [Background] Morote Robles J, Lorente JA, Reig C, Lopez Pacios MA, de Torres JA, Soler Rosello A. [The clinical and prognostic value of inversion of the PSA/PAP ratio in prostatic cancer]. Actas Urol Esp. 1994 May;18(5):559-61. Spanish. PMID 7521563